CLINICAL TRIAL: NCT03221543
Title: The Role of Pre-Surgical Metabolic Testing for Procedure Selection in Bariatric Surgery
Brief Title: Resting Metabolic Rate Testing in Bariatric Surgery Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In this study, there is 1 year of active subject participation and long-term follow-up data collected at year 5. Since study objectives were met with active subject data, the study team will not be collecting long-term data at year 5.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 017-125
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Weight Loss; Bariatric Surgery Candidate
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Resting Metabolic Rate Testing (Experimental): All subjects will have the resting metabolic rate test. The ReeVue Indirect Calorimeter from Korr Medical will be used to obtain the resting metabolic rate.
  Interventions: Device: ReeVue Indirect Calorimeter

INTERVENTIONS:
Device: ReeVue Indirect Calorimeter — The ReeVue Indirect Calorimeter will be used in this study to measure the resting metabolic rate. The test takes approximately ten minutes to complete. The subject should prepare for the test by avoiding stimulants and exercise on the day of the test, as well as eating meals four hours before the test. The subject will be seated during the test. They will be given a nose clip that looks like a clothes pin to be placed on their nose. A plastic mouth piece that allows all of the air they breathe to come in through the top of the mouth piece and the air they breathe out to go into the ReeVue Calorimeter will also be provided. The subject will remain in this position for ten minutes until the testing is complete.

SUMMARY:
This study evaluates if measuring resting metabolic rate (the number of calories the body burns at rest) before surgery can help predict successful weight loss after surgery.

DETAILED DESCRIPTION:
This is a prospective study enrolling patients from the Baylor Weight Loss Surgery Center who have met all of the requirements to proceed with primary bariatric surgery. Patients will undergo pre-operative and post-operative metabolic testing (6 months, and 1 year after surgery) using a portable calorimeter with eventual follow up of medical record at 5 years. Data from up to 50 patients will be collected. The main objectives are to examine if the pre-operative resting metabolic rate can accurately predict successful weight loss after bariatric surgery and if it can be used to guide the selection of the type of bariatric surgery that would be most successful for the patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for a primary bariatric surgery
* 18 years of age to no upper limit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Examine percent total weight loss | 1 year
  Weigh subjects using a scale

SECONDARY OUTCOMES:
Change in resting metabolic rate | 1 year
  Obtain resting metabolic rate using the Reevue Indirect Calorimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Weight Loss Surgery Center, Dallas, Texas, United States